CLINICAL TRIAL: NCT03481816
Title: Treatment of Patients With Castration Resistant Prostate Cancer Using a Multi-Targeted Recombinant Ad5 PSA/MUC1/Brachyury Based Immunotherapy Vaccines
Brief Title: Treatment of Castration Resistant Prostate Cancer Using Multi-Targeted Recombinant Ad5 PSA/MUC1/Brachyury Based Immunotherapy Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marijo Bilusic, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 180073; 18-C-0073
Record Dates: First submitted 2018-03-28; First posted 2018-03-29 (Actual); Results first posted 2020-12-22 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Prostatic Neoplasms; Prostatic Cancer
Keywords: mCRPC; Therapeutic Cancer Vaccines; ETBX-071; ETBX-061; ETBX-051
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1/Dose De-Escalation (Experimental): Subjects enrolled to dose de-escalation cohorts.
  Interventions: Biological: ETBX-071; adenoviral PSA vaccine; Biological: ETBX-061; adenoviral MUC1 vaccine; Biological: ETBX-051; adenoviral brachyury vaccine
- Arm 2/Dose expansion (Experimental): Subjects enrolled at the maximum tolerated dose (MTD) after the MTD is established.
  Interventions: Biological: ETBX-071; adenoviral PSA vaccine; Biological: ETBX-061; adenoviral MUC1 vaccine; Biological: ETBX-051; adenoviral brachyury vaccine

INTERVENTIONS:
Biological: ETBX-071; adenoviral PSA vaccine — 5 x 10 to the eleventh power VP (standard dose), 1 x 10 to the eleventh power VP (DL-1), or 5 x 10 to the tenth power VP (DL-2) subcutaneous injection every 3 weeks for 3 immunizations.
Biological: ETBX-061; adenoviral MUC1 vaccine — 5 x 10 to the eleventh power VP (standard dose), 1 x 10 to the eleventh power VP (DL-1), or 5 x 10 to the tenth power VP (DL-2) subcutaneous injection every 3 weeks for 3 immunizations.
Biological: ETBX-051; adenoviral brachyury vaccine — 5 x 10 to the eleventh power VP (standard dose), 1 x 10 to the eleventh power VP (DL-1), or 5 x 10 to the tenth power VP (DL-2) subcutaneous injection every 3 weeks for 3 immunizations.

SUMMARY:
Background:

Metastatic castration resistant prostate cancer (mCRPC) keeps growing even when the amount of testosterone in the body is reduced to very low levels. mCRPC is incurable. Researchers want to develop vaccines to teach the immune system to target and kill cancer cells. They want to test three of these vaccines (ETBX-071, ETBX-061, and ETBX-051) against mCRPC.

Objective:

To test the safety of combination ETBX-071, ETBX-061, and ETBX-051 and to study their effects on the immune system.

Eligibility:

People ages 18 and older with mCRPC that has not responded to standard therapies

Design:

Participants will be screened with:

Medical history

Physical exam

Blood, urine, and heart tests

Computed tomography (CT) or magnetic resonance imaging (MRI) scans

Bone scan

Participants will get the vaccines as shots under the skin every 3 weeks for 3 doses. They may then have the shots every 8 weeks for up to 1 year.

Participants will keep a diary to record any symptoms from the vaccines.

Participants will have blood tests each time they get the vaccines. They will also have scans and other tests to measure the effect the vaccines have on their tumors.

Participants will have a visit within 28 days after their last treatment. This includes a physical exam and blood and urine tests.

Participants will then be contacted by phone every 3 months for the first year, every 6 months for the next 2 years, and every 12 months for another 2 years.

Participants will be asked to join a long-term follow up study.

DETAILED DESCRIPTION:
Background:

* The overall goal of the current project is to expand our immunotherapeutic approach for the treatment of prostate cancer employing a multi-targeted approach.
* Therapeutic cancer vaccines targeting overexpressed proteins offer a potential method to activate T cells against tumors.
* A novel adenovirus based vaccines targeting three (3) human tumor associated antigens (TAA), Prostate specific antigen (PSA), Mucin 1 (MUC1), and brachyury, respectively have demonstrated anti-tumor cytolytic T cell responses in pre-clinical animal models of cancer.

Objectives:

-To determine the overall safety and recommended phase 2 dose of a combination of three immunotherapeutic vaccines (ETBX-071, ETBX-061, and ETBX-051) when administered subcutaneously (SC) to subjects with metastatic castration resistant prostate cancer

Eligibility:

* Subjects age 18 and older with cytologically or histologically confirmed prostate cancer for which no curative standard approved therapy is available.
* Metastatic Castration Resistant Prostate Cancer (mCRPC) patients with rising PSA or progressive disease despite castration levels of testosterone.
* Prior treatment with immunotherapy hormonal therapy, radiotherapy, chemotherapy, and/or other experimental therapy is allowed.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1
* Adequate organ and bone marrow function
* Subjects with a history of autoimmune disease (active or past) and subjects requiring systemic steroids are not eligible (physiologic doses of steroids for steroid replacement as well as nasal, topical and inhaled steroids are allowed). Autoimmune-related thyroid disease, type I diabetes and vitiligo are permitted if the condition is well controlled.

Design:

* This is a Phase I trial in subjects with mCRPC. A combination of three therapeutic vaccines (ETBX-071, ETBX-061, and ETBX-051) which use the same modified Adenovirus vector backbone, separately encoding three well studied TAA,PSA, MUC1, and brachyury, respectively) will be assessed. The vaccines will be tested at standard dose levels, with a dose de-escalation (if required) design employed. The dose level of each vaccine tested will be 5x10 to the eleventh power VP. This dose has been found in a prior phase 1 testing of a similar vaccine Ad5 [E1-, E2b-]-carcinoembryonic antigen (CEA)(6D) (ETBX-011) to be well tolerated (with no dose-limiting toxicities (DLTs) or related serious adverse events(SAEs), and be optimal for induction of immune responses.
* Up to six patients will be enrolled at dose level 1. If less than or equal to 1 of 6 patients experience a DLT, an initiation of the dose expansion phase will occur. If more than or equal to 2 of 6 experience DLT at dose level 1, then dose de-escalation will occur. Up to six patients will be enrolled at the lower dose level (-1) (1x10 to the eleventh power VP). If less than or equal to 1 of 6 patients experience a DLT, then the maximum tolerated (MTD) will be declared at this dose, and initiation of the dose expansion phase will occur. If more than or equal to 2 of 6 experience DLT at dose level -1, then a further dose de-escalation will occur. Up to six patients will be enrolled at the lower dose level (-2) (5x10 to the tenth power VP). If less than or equal to 1 of 6 patients experience a DLT, then the maximum tolerated (MTD) will be declared at this dose, and initiation of the dose expansion phase will occur. If more than or equal to 2 of 6 experience DLT at dose level -2, then the study will be stopped.
* A dose expansion phase of study will be enrolled after the MTD of the vaccines have been determined. An additional 12 subjects will be enrolled in the dose expansion component of the trial, for a total of 18 subjects at the MTD.
* The ETBX-051, ETBX-61 and ETBX-71 vaccines will be administered subcutaneously (SC) at separate injection sites (proximal limb, preferably the thigh), will be administered SC every 3 weeks for 3 doses (dose de-escalation cohorts) followed by boosts every 8 weeks for 1 year (only patients enrolled in dose expansion cohort).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age more than or equal to 18 years (male).
* Ability to understand and provide signed informed consent that fulfills Institutional Review Board (IRB)s guidelines.
* Cytologically or histologically confirmed prostate cancer for which no curative standard approved therapy is available by either the Laboratory of Pathology at the National Institutes of Health (NIH) Clinical Center or Walter Reed National Military Medical Center at Bethesda prior to starting this study. If no pathologic specimen is available, patients may enroll with a pathologists report showing a histological diagnosis of prostate cancer and a clinical course consistent with the disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Subjects who have received prior prostate specific antigen (PSA), mucin1 (MUC1), and/or brachyury-targeted immunotherapy (e.g. vaccine) are eligible for this trial if this treatment was discontinued at least 3 months prior to enrollment.
* Resolution of all toxic side effects of prior chemotherapy, radiotherapy, or surgical procedures to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade less than or equal to1.
* Adequate hematologic function at screening, as follows:
* Absolute neutrophil count (ANC) greater than or equal to x 10 to the ninth power/L
* Hemoglobin more than or equa to 9 g/dL
* Platelets more than or equal to 75,000/microliter.
* Prothrombin (PT)-international normalized ratio (INR) < 1.5.
* Partial thromboplastin time (PTT) < 1.5 x upper limit of normal (ULN).
* Adequate renal and hepatic function at screening, as follows:

  --Serum creatine less than or equal to 1.5x upper limit of normal (ULN) OR creatinine clearance (CrCl) more than or equal to 40mL/min (if using the Cockcroft-Gault formula below):
  1. Female CrCl = [(140 - age in years) x weight in kg x 0.85] / [72 x serum creatinine in mg/dL]
  2. Male CrCl = [(140 - age in years) x weight in kg x1.00] / [72 x serum creatinine in mg/dL]
* Total bilirubin less than or equal to 1.5 x ULN OR in subjects with Gilberts syndrome, a total bilirubin less than or equal to x ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 2.5 x ULN, unless liver metastasis are present, then values must be less than or equal to 5 x ULN)
* The effects of ETBX-051, ETBX-061 and ETBX-071 vaccines on the developing human fetus are unknown. For this reason subjects must agree to use a condom and acceptable contraceptive method with their partner during the study and for one month after the last dose of vaccines.
* Ability to attend required study visits and return for adequate follow up, as required by this protocol.
* Castrate testosterone level (<50ng/dl or 1.7nmol /L)
* Metastatic disease documented by at least one of the following:
* Metastatic bone disease on an imaging study, or
* Soft tissue disease documented by computed tomography (CT)/magnetic resonance imaging (MRI)
* Progressive disease at study entry defined as one or more of the following criteria occurring in the setting of castrate levels of testosterone:
* Radiographic progression defined as any new or enlarging bone lesions or growing lymph node disease, consistent with prostate cancer

OR

* PSA progression defined by sequence of rising values separated by >1 week (2 separate increasing values over a minimum of 2ng/ml (Prostrate Cancer Working Group 2 (PCWG2) PSA eligibility criteria). If patients had been on flutamide, PSA progression is documented 4 weeks or more after withdrawal. For patients on bicalutamide or nilutamide disease progression is documented 6 or more weeks after withdrawal. The requirement for a 4-6 week withdrawal period following discontinuation of flutamide, nilutamide or bicalutamide only applies to patients who have been on these drugs for at least the prior 6 months. For all other patients, they must stop bicalutamide, nilutamide or flutamide the day prior to enrollment.
* Patients must agree to continue to continuation of androgen deprivation therapy (ADT) with a gonadotropin-releasing hormone analogue/antagonist or bilateral orchiectomy
* Prior treatment with immunotherapy, hormonal therapy, radium 223, chemotherapy and/or other experimental therapy is allowed.

EXCLUSION CRITERIA:

* Treatment with an investigational drug study within 28 days of before starting on study treatment.
* Subjects with concurrent cytotoxic chemotherapy or radiation therapy. There must be at least 28 days between any other prior chemotherapy (or radiotherapy) and study treatment. Prior antibody therapy must be discontinued 8 weeks prior to start of study treatment. Prior hormonal therapy can be discontinued 24 hours prior to start of study treatment.
* Any prior PSA, MUC1, and/or brachyury-targeted immunotherapy (e.g., vaccine) must have been discontinued at least 12 weeks before initiation of study treatment. Subjects must have recovered from all acute toxicities from prior treatment prior to screening for this study.
* Prior treatment with Adenovirus-Based vectors immunotherapy
* Known active brain or central nervous system metastasis, or seizures requiring anticonvulsant treatment, cerebrovascular accident, or transient ischemic attack (< 6 months prior to enrollment).
* Subjects with a history of autoimmune disease (active or past), such as but not restricted to inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis. Autoimmune-related thyroid disease, type I diabetes and vitiligo are permitted if the condition is well controlled.
* Subjects with serious intercurrent chronic or acute illness, such as cardiac or pulmonary disease, hepatic disease, or other illness considered by the Investigator as high risk for investigational drug treatment.
* Subjects with a history of heart disease, such as congestive heart failure (class II, III, or IV defined by the New York Heart Association functional classification), history of unstable or poorly controlled angina, or history (< 1 year prior to enrollment) of ventricular arrhythmia.
* Subjects with a medical or psychological impediment that would impair the ability of the subject to receive therapy per protocol or impact ability to comply with the protocol or protocol-required visits and procedures.
* Presence of a known active acute or chronic infection, including human immunodeficiency virus (HIV, as determined by enzyme-linked immunosorbent assay [ELISA] and confirmed by western blot) and hepatitis B and hepatitis C virus (HBV/HCV, as determined by Hepatitis B surface antigen (HBsAg) and hepatitis C serology).
* Subjects on systemic intravenous or oral steroid therapy (or other immunosuppressive, such as azathioprine or cyclosporin A) are excluded on the basis of potential immune suppression. Subjects must have had at least 6 weeks of discontinuation of any steroid therapy (except that used as premedication for chemotherapy or contrast-enhanced studies) prior to enrollment. Physiologic (replacement) doses of steroids as well as nasal, topical or inhaled steroids are allowed.
* Subjects with known allergy or hypersensitivity to any component of the investigational product will be excluded.
* Subjects with acute or chronic skin disorders that will interfere with injection into the skin of the extremities or subsequent assessment of potential skin reactions will be excluded.
* Subjects vaccinated with a live (attenuated) vaccine (e.g., FluMist) or a killed (inactivated)/subunit vaccine (e.g., PNEUMOVAX, Fluzone) within 28 days or 14 days, respectively, of the first planned dose of ETBX vaccine.
* Patients with second malignancy within 3 years of enrollment; Patients curatively treated non-melanoma skin cancers or carcinoma in situ of the bladder, are not excluded.
* Use of herbal products that may decrease PSA levels (e.g. saw palmetto)
* Patients who have received radiation therapy, radionuclide therapy or undergone surgery within certain duration (4 weeks) of enrollment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marijo Bilusic, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bilusic M, McMahon S, Madan RA, Karzai F, Tsai YT, Donahue RN, Palena C, Jochems C, Marte JL, Floudas C, Strauss J, Redman J, Abdul Sater H, Rabizadeh S, Soon-Shiong P, Schlom J, Gulley JL. Phase I study of a multitargeted recombinant Ad5 PSA/MUC-1/brachyury-based immunotherapy vaccine in patients with metastatic castration-resistant prostate cancer (mCRPC). J Immunother Cancer. 2021 Mar;9(3):e002374. doi: 10.1136/jitc-2021-002374. PMID 33762322
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0073.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1/Dose De-escalation: Subjects enrolled to dose de-escalation cohorts. We did not need to dose de-escalate since none of patient's had dose limiting toxicity (DLT) so all patients received planned higher starting dose.
  ETBX-071; adenoviral PSA vaccine: 5 x 10 to the eleventh power VP (standard dose), 1 x 10 to the eleventh power VP (DL-1), or 5 x 10 to the tenth power VP (DL-2) subcutaneous injection every 3 weeks for 3 immunizations.
  ETBX-061; adenoviral MUC1 vaccine: 5 x 10 to the eleventh power VP (standard dose), 1 x 10 to the eleventh power VP (DL-1), or 5 x 10 to the tenth power VP (DL-2) subcutaneous injection every 3 weeks for 3 immunizations.
  ETBX-051; adenoviral brachyury vaccine: 5 x 10 to the eleventh power VP (standard dose), 1 x 10 to the eleventh power VP (DL-1), or 5 x 10 to the tenth power VP (DL-2) subcutaneous injection every 3 weeks for 3 immunizations.
Period: Starting Dose
Arm/Group | Arm 1/Dose De-escalation | Arm 2/Dose Expansion
Started | 6 | 0
Completed | 5 | 0
Not Completed | 1 | 0
Not completed — Refused further vaccines after 1 dose | 1 | 0
Period: Dose Expansion
Arm/Group | Arm 1/Dose De-escalation | Arm 2/Dose Expansion
Started | 0 | 12
Completed | 0 | 0
Not Completed | 0 | 12
Not completed — Off treatment due to progressive disease | 0 | 5
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Physician Decision | 0 | 5

BASELINE CHARACTERISTICS:
Population: We did not need to dose de-escalate since none of patient's had dose limiting toxicity (DLT) so all patients received planned higher starting dose in Arm 1/Dose De-escalation Arm/Group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1/Dose De-Escalation | Arm 2/Dose Expansion | Total
Number analyzed (Participants) | 6 | 12 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 5 | 10 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.62 (8.6) | 72.58 (9.23) | 71.60 (8.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 12 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 12 | 17
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 4 | 11 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 12 | 18
Median Baseline Prostate-Specific Antigen (PSA) [Median (Full Range); unit: ng/mL] | 46.92 [8.01 to 1006] | 14.55 [0.65 to 605] | 25.58 [0.65 to 1006]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities
Description: A dose-limiting toxicity is defined as occurring within 28 days after the first vaccine administration and meeting on of these criteria: Any Grade 3 or greater toxicity or any Grade 2 or higher autoimmune reaction as defined by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0; or generalized erythroderma or macular or papular rash.
Time Frame: 4 weeks after receiving the first vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1/Dose De-Escalation | Arm 2/Dose Expansion
Number analyzed (Participants) | 6 | 12
Participants | 0 | 0

2. Primary Outcome: Recommended Phase 2 Dose
Description: RP2D is the maximum tolerated dose declared after ≤1 of 6 participants experience a dose-limiting toxicity within the first 4 weeks.
Time Frame: Within the first 4 weeks after drug is administered.
Measure: Number; unit: viral particles
Arm/Group | Arm 1/Dose De-Escalation
Number analyzed (Participants) | 6
viral particles | 500000000000

3. Secondary Outcome: Percentage of Participants With an Objective Response
Description: ORR is the percentage of subjects who experience partial response (PR) or complete response (CR) measured by the Response Evaluation Criteria in Solid Tumors (RECIST) at any time point during the treatment period. PR is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Time Frame: Objective response at any time point during treatment on study up to 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1/Dose De-Escalation | Arm 2/Dose Expansion
Number analyzed (Participants) | 6 | 12
percentage of participants
  Partial Response | 0 | 8.3
  Complete Response | 0 | 0

4. Secondary Outcome: Percentage of Participants With a Disease Control Rate (DCR) Lasting for at Least 6 Months
Description: DCR is the percentage of subjects who experience partial response (PR), complete response (CR), or stable disease (SD) lasting for at least 6 months. Response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST)v1. PR is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum of diameters while on study. Progressive disease is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions.
Time Frame: 6 months post treatment
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1/Dose De-Escalation | Arm 2/Dose Expansion
Number analyzed (Participants) | 6 | 12
percentage of participants
  Partial Response | 0 | 8.3
  Complete Response | 0 | 0
  Stable Disease | 0 | 41.6

5. Secondary Outcome: Duration of Response
Description: Duration of response is the time from when measurement criteria for Partial Response (PR) or Complete Response (CR) are met until disease recurrence or progression per dose cohort. Response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST)v1. PR is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progressions.
Time Frame: Time from recorded partial response until development of progressive disease. This was accessed every 3 weeks for the first 3 doses and then every 8 weeks up to 1 year (Arm 2)
Population: Per protocol, this outcome measure was pre-specified to be performed in Arm 2 only.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Arm 2/Dose Expansion
Number analyzed (Participants) | 1
Weeks | 16 [NA to NA] — The full range cannot be calculated because we need at least two values. 1/12 participants had a response and was analyzed.

6. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is the time from the date of first treatment to the date of disease progression or death (any cause) whichever occurs first per dose cohort. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST)v1. Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progressions.
Time Frame: This was accessed every 3 weeks for the first 3 doses, then every 8 weeks up to 1 year (Arm 2).
Population: Per protocol, this outcome measure was pre-specified to be performed in Arm 2 only.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Arm 2/Dose Expansion
Number analyzed (Participants) | 12
Weeks | 22 [19.1 to 34]

7. Secondary Outcome: Overall Survival (OS)
Description: OS is the time from the date of first treatment to the date of death (any cause).
Time Frame: Every 3 weeks for the first 3 doses, then every 8 weeks up to 1 year then every 3 months for 12 months and then approximately every 6 months every 6 months for 24 months and then every 12 months thereafter for another 24 months.
Population: Median OS not reached. Per protocol we have to assess Overall survival (OS) - the time from the date of first treatment to the date of death (any cause) per dose cohort and overall.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Arm 1/Dose De-Escalation | Arm 2/Dose Expansion
Number analyzed (Participants) | 6 | 12
Weeks | 12.2 [3.3 to NA] — There is no upper end with "not estimable". | NA [NA to NA] — Median OS not reached as no events occurred (all patients are alive)

8. Secondary Outcome: Percentage of Overall Survival (OS) Probability at 12 Months and 24 Months
Description: Probability of being alive at 12 Months and 24 Months after first vaccine.
Time Frame: 12 and 24 months after first treatment
Measure: Median (95% Confidence Interval); unit: Percentage of probability
Arm/Group | Arm 1/Dose De-Escalation | Arm 2/Dose Expansion
Number analyzed (Participants) | 6 | 12
Percentage of probability
  12 Months | 50.0 [11.1 to 80.4] | 100 [100 to 100]
  24 Months | 33.3 [4.6 to 67.6] | 100 [100 to 100]

9. Secondary Outcome: Prostate-Specific Antigen Doubling Time (PSA DT) at Week 14 and End of Study
Description: PSA DT in participants with advanced cancer treated with the ETBX-071, ETBX-061, and ETBX-051 vaccines were determined using a nomogram to find detectable PSA.
Time Frame: PSA DT was done once at week 14 and the second time at the end of study (any time point within a year while on study when they met criteria for progression)
Measure: Median (Standard Deviation); unit: Months
Arm/Group | Arm 1/Dose De-Escalation | Arm 2/Dose Expansion
Number analyzed (Participants) | 6 | 12
Months
  Week 14 | NA (NA) — The first 6 patients completed study after 6 weeks, therefore we did not calculate PSA DT at end of study treatment). | 2.4 (23.9)
  End of Study | NA (NA) — The first 6 patients completed study after 6 weeks, therefore we did not calculate PSA DT at end of study treatment). | 4.3 (4.97)

10. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 8 months and 30 days for the Arm 1/Dose De-Escalation group, and 10 months and 25 days for the Arm 2/Dose Expansion group.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1/Dose De-Escalation | Arm 2/Dose Expansion
Number analyzed (Participants) | 6 | 12
Participants | 6 | 12

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 8 months and 30 days for the Arm 1/Dose De-Escalation group, and 10 months and 25 days for the Arm 2/Dose Expansion group.
Arm/Group | Arm 1/Dose De-Escalation | Arm 2/Dose Expansion
All-Cause Mortality (participants affected / at risk) | 4/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/12
Other Adverse Events (participants affected / at risk) | 6/6 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1/Dose De-Escalation (N=6) | Arm 2/Dose Expansion (N=12)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1/Dose De-Escalation (N=6) | Arm 2/Dose Expansion (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 4 (4) | 3 (3)
Fever (General disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 3 (3) | 7 (8)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Injection site reaction (Injury, poisoning and procedural complications) | 6 (7) | 11 (22)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2)
Weight loss (Investigations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT03481816/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT03481816/ICF_001.pdf